CLINICAL TRIAL: NCT01733199
Title: Behavioural Addictions Occurring During a Dopaminergic Treatment Prescribe Under Parkinson's Disease: Study of the Psychopathological, Neurological, Pharmacokinetic and Genetic Profiles.
Acronym: PARKADD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC12_0059
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Parkinson's Disease; Secondary Behavioural Addiction
Keywords: Parkinson's disease; Behavioural addictions; Pathological gambling; Dopamine agonist; Dopamine dysregulation syndrome; Pharmacokinetic; Pramipexole
MeSH Terms: conditions — Parkinson Disease; Gambling | interventions — Surveys and Questionnaires

ARMS (3):
- BA- (Experimental): Patient with no secondary behavioural addiction
  Interventions: Other: questionnaires
- BA+/DDS- (Experimental): Patients with secondary behavioural addiction, without dopamine dysregulation syndrome
  Interventions: Other: questionnaires
- BA+/DDS+ (Experimental): Patients with secondary behavioural addiction and dopamine dysregulation syndrome
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Summons of patients and filling questionnaire.

SUMMARY:
This study is composed of a main study and an ancillary one. The objective of the main study is to define, on the psychopathological, neurological, pharmacokinetic and genetic plan, the predictive factors for developing a behavioural addiction (BA) secondarily to the dopaminergic treatment, associated or not to a dopamine dysregulation syndrome (DDS), in patients with Parkinson's disease.

3 particular profiles of patients will be established:

* BA- : no secondary behavioural addiction
* BA+/DDS-: secondary behavioural addiction, without dopamine dysregulation syndrome
* BA+/DDS+: secondary behavioural addiction, with dopamine dysregulation syndrome

We wish in particular:

* To differentiate, among the BA+ subjects, those for who is a DDS from those for who we can evoke a side effect of the dopaminergic treatment
* To demonstrate that the BA+/DDS- subjects present pharmacokinetic particularities causing the occurrence of the BA.
* To clarify the possible relationship between the dosage and the pharmacodynamics of the treatment (especially that of pramipexole) in one hand, and the developing of BA in the other hand.
* Demonstrate that the subjects BA + / DDS- are individually genetic vulnerability (related to the dopamine system), originally from the occurrence of the BA.

This study has several levels of evaluation, we chose describe the methodology of the study in 3 axis : Psychopathology axis, Neurological axis and pharmacokinetic axis.

The pharmacokinetic aspects will be studied only on a part of the sample, in an ancillary study centered on the pharmacokinetic of the pramipexole (in its immediate release form).

DETAILED DESCRIPTION:
This is a monocentric study with a recruitment period comprised between October 2012 and April 2016. The recruitment occurs during the consultations in the service of neurology. If the subjects are eligible, the study is proposed to them, and an evaluation is fixed in the next days. This evaluation consists in an individual face-to-face interview based on standardized and semi-structured questionnaires, during approximately one and a half hour. It's focused on the different characteristics of Parkinson's disease, and on psychiatric and addictive co morbidities. The evaluation is completed by a set of self-administered questionnaires focused on impulsivity and Attention Deficit Hyperactivity Disorder (ADHD).

For the 80 patients participated to the ancillary study only, a blood sample will be realized when the patient will arrived, just before the intake of his treatment (to obtain the residual plasmatic concentration). A second sample will be realized at a different time for each patient, to cover the entirety of the kinetic between 2 intakes of pramipexole (immediate release form) via the entire sample. The second blood sample will be realized four hours after the first one at the most. After this second sample, the patient will have completed his participation to the study.

Secondly, monitoring including a self-questionnaire booklet and a saliva sample will be offered to all patients who completed the initial visit.

ELIGIBILITY:
Main study

Inclusion criteria:

* To be 18 years old or more (both genders)
* To have idiopathic Parkinson's disease, without important cognitive troubles, treated by usually prescribed drugs
* To have a treatment established since 6 months at least

Exclusion criteria:

* To be under tutelage (a French protecting measure for persons with altered judgement)
* To have a secondary Parkinson's disease
* To have received a chirurgical treatment for Parkinson's disease
* To present obvious cognitive disturbances

Ancillary study (pharmacokinetic axis) :

Inclusion criteria:

* The same as the main study
* To have a treatment by pramipexole in the immediate release form

Exclusion criteria:

* The same as the main study
* Association of the pramipexole with others molecules
* To use to have a behavioural addiction resolved by a diminution of the dosage before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Psychopathological axis : score of sensation seeking (S Score) of the impulsivity questionnaire "UPPS"
  This choice is founded on the fact that patients suffering of DDS are described as being impulsive, misusing their anti-parkinsonism treatment in the purpose of stimulate themselves, suggesting they have a high level of sensation and novelty seeking.
Pharmacological axis : Area under the curve of the pramipexole concentration
  Area under the curve of the pramipexole concentration in function of the time between 2 intakes of pramipexole.
Neurological axis : Unified Parkinson's Disease Rating Scale (UPDRS) III score
  UPDRS III score, with axial under-score in ON and OFF DOPA (Parkinson's disease severity)
Genetic axis : distribution of allele frequencies and genotypic
  Distribution of allele frequencies and genotypic

SECONDARY OUTCOMES:
Treatments except the anti-parkinsonism ones
  Psychopathological axis
drug misuse
  Psychopathological axis
addiction and punding antecedents
  Psychopathological axis
ADHD antecedents
  Psychopathological axis
impulsivity profile
  Psychopathological axis
Age of onset of the Parkinson's disease
  Neurological axis
stage and form of the Parkinson's disease
  Neurological axis included dyskinesia and involuntary abnormal movements
time course of Parkinson's disease
  Neurological axis
family history of Parkinson's disease
  Neurological axis
anti-parkinsonism treatments
  Neurological axis
Residual plasmatic concentration of the pramipexole
  Pharmacological axis The data of the pharmacological axis are measured after analyzes of the blood samples collected in that evaluation, only for the 80 patients participated to the ancillary study.
median pharmacokinetic parameters of pramipexole
  Pharmacological axis The data of the pharmacological axis are measured after analyzes of the blood samples collected in that evaluation, only for the 80 patients participated to the ancillary study.
study of the hepatic and renal functions
  Pharmacological axis The data of the pharmacological axis are measured after analyzes of the blood samples collected in that evaluation, only for the 80 patients participated to the ancillary study.
Physiopathological covariates
  Pharmacological axis age, gender, weight, creatinine and prothrombin rates The data of the pharmacological axis are measured after analyzes of the blood samples collected in that evaluation, only for the 80 patients participated to the ancillary study.

CONTACTS AND LOCATIONS:
Overall Officials: Marie GRALL-BRONNEC, Principal Investigator — Nantes UH
Locations (1):
- Nantes University Hospital, Nantes, France